CLINICAL TRIAL: NCT03459235
Title: Assessment of Functional Digestive and Genitourinary Outcomes in Patients With Rectal Cancer Living After 2 Years Without Recurrence. Population Study. (Rectqol)
Brief Title: Assessment of Functional Digestive and Genitourinary Outcomes in Patients With Rectal Cancer.
Acronym: Rectqol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017 - A02645-48
Record Dates: First submitted 2017-12-22; First posted 2018-03-08 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-03

CONDITIONS: Rectal Cancer; Surgery
Keywords: rectal cancer; proctectomy; digestive sequelae; quality of life; Urinary and Sexual sequelae
MeSH Terms: conditions — Rectal Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- population from registry data (Experimental): the intervention involves completing several quality of life questionnaires validated in the medical literature (LARS score, FSFI, USP, IIEF, IPPS, QLQ C-30, QLQ-CR29)
  Interventions: Other: quality of life

INTERVENTIONS:
Other: quality of life — Assessment of the impact of digestive sequelae (LARS score) and genitourinary sequelae (score IPSS, USP, FSFI et IIEF) in Patients With Rectal Cancer using validated questionnaires on quality of life (EORTC QLQ-C30 et QLQ-CR 29).

SUMMARY:
Total mesorectal excision and neoadjuvant radio-chemotherapy have revolutionized the management of rectal cancer allowing an increase in survival (between 55 and 68% at 5 years) and allowing a decrease of local recurrence (under 10%) and allowing to push the limits of sphinctyer saving procedures.

Parallel to the oncological findings, evaluating quality of life and functionnals sequelae has become a priority as highlighted by the second axis of "plan cancer 2014-2019".

The prevalence of digestive functional sequelae decrease during the first two years after surgery. However, these results are difficult to analyse due to the heterogeneity of used scores in medical litterature. The low anterior resection syndrom associate poly-exoneration, gas and / or stool incontinence, urgency and stool splitting.

The score of low anterior resection " LARS score " validated in Danemark in 2012 allow us to understand the complexity of these sequelae and to measure their impact on the quality of life of patients, that's why he is currently recommended.

In the long term, almost two out of three patients suffer from this syndrom, with half of the patients in a severe form.

However, its prevalence and severity are often underestimated by practitioners. It leads to inappropriate therapeutic measures. The aim of this study is to evaluate the impact of digestive and genito-urinary sequelae on quality of life from validated scores in patients operated curatively of rectal cancer using a population study.

This study should include 676 patients with rectal cancer treated in calvados and alive at 2 years of their proctectomy without local or general recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for a rectal adénocarcinoma with a curative aim with or without neo-adjuvating treatment in Calvados between January 1st, 2007 (date of recommendations for clinical practise) and december 31 th, 2014.
* Patients having their main address in the Calvados (at the time of diagnosis) and recorded in the register of digestive tumors of the Calvados.
* patients alive on first of january 2018 without local recurrence nor global recurrence
* patients able to understant a validated questionnaire.

Exclusion Criteria:

* Dead patients
* patients with cancer recurrence
* Patient with severe cognitive disorders (confusions) preventing the good understanding of questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-06-15 (Estimated)

PRIMARY OUTCOMES:
assessment of digestive sequelae in patients operated for a rectal cancer (rectal resection) | more than 2 years after rectal resection
  score used : LARS score (for men and women). 5 questions about the low anterior resection syndrom. Scale between 0 and 42 points. Better outcome is 0 and worse is 42.
assessment of global quality of life in patients operated for a rectal cancer (rectal resection) | more than 2 years after rectal resection
  Score used : EORTC - QLQ C-30 - European Organization for research and treatment of cancer Quality of Life Questionnaire Core 30 (for men and women). It is a scale to evaluate the generic quality of life after cancer. There are 30 questions : 28 questions with 4 possible answers from 1 to 4 and 2 questions to evaluate the physical state and global quality of life with answers between 1 and 7. For each answer, 1 is the worst outcome and 4 is the best except for the 2 last questions where 7 is the best outcome. Minimum (worst outcome) is 30 and best outcome is 126. The total is reported to a score of 100 points which is the best outcome.
assessment of specific quality of life in patients operated for a rectal cancer (rectal resection) | more than 2 years after rectal resection
  score used : EORTC - QLQ CR 29 European Organization for research and treatment of cancer Quality of Life Questionnaire Colorecatl module 29 (for men and women). This score is used in patients undergoing treatment for colorectal cancer. There are 29 questions with 4 possible answers (between 1 and 4 points). Best outcome is 4 for each question. Worst outcome is 1 for each question. Minimum (worst outcome) is 29 and best outcome is 116. The total is reported to a score of 100 points which is the best outcome.
assessment of quality of life of patients operated for a rectal cancer (rectal resection) - urinary sequelae (for women) | more than 2 years after rectal resection
  score used : Urinary Symptom Profile : USP (for women). This scale is used to evaluate urinary symptoms. 1 question to evaluate stress urinary incontinence (between 0 and 9 points). 9 points is the worts outcome. 7 questions to evaluate overactive bladder symtoms (between 0 points and 21). 21 points is the worst outcome. 3 questions to evaluate low stream symtoms (between 0 and 9 points). 9 points is the worst outcome.
  Global score is between 0 and 39 points. 39 points is the worst outcome and 0 points the best outcome.
assessment of quality of life of patients operated for a rectal cancer (rectal resection) - urinary sequelae (for men) | more than 2 years after rectal resection
  score used : International Prostate Score Symptom : IPSS (for men). There are 7 questions with 5 possible answers (between 0 (best outcome) and 5 (worst outcome)). And one additionnal question to evaluate quality of life due to urinary symptom with 7 possible answers from 0 (best outcome) to 6 (worst outcome). for the seven first questions : best outcome is 0 and worst outcome is 35. For the last question 0 is the best and 6 is the worst outcome).
assessment of quality of life of patients operated for a rectal cancer (rectal resection) - Sexual sequelae (for women) | more than 2 years after rectal resection
  score used : Female Sexual Functionnal index : FSFI (for women). 19 questions on sexual sequelae in this questionnaire. Worst outcome is 2 and best outcome is 95 points.
assessment of quality of life of patients operated for a rectal cancer (rectal resection) - Sexual sequelae (for men) | more than 2 years after rectal resection
  score used : International Index for Erectile Function 5 : IIEF 5 (for men). 5 questions for sexual quality of life in males. Each questions have 5 answers. 5 points is the best outcome for each question. Minimal score is 1 and best score (best outcome) is 25.

CONTACTS AND LOCATIONS:
Locations (1):
- François baclesse Center - U1086 - Anticipe, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alves A. [Recommendations for clinical practice. Therapeutic choices for rectal cancer. How can we reduce therapeutic sequelae and preserve quality of life?]. Gastroenterol Clin Biol. 2007 Jan;31 Spec No 1:1S52-62, 1S95-7. No abstract available. French. PMID 17569477
- [Result] Abdelli A, Tillou X, Alves A, Menahem B. Genito-urinary sequelae after carcinological rectal resection: What to tell patients in 2017. J Visc Surg. 2017 Apr;154(2):93-104. doi: 10.1016/j.jviscsurg.2016.10.002. Epub 2017 Feb 1. PMID 28161008
- [Result] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Derived] Eid Y, Bouvier V, Menahem B, Thobie A, Dolet N, Finochi M, Renier M, Gardy J, Launoy G, Dejardin O, Morello R, Alves A; Rectqol Group. Digestive and genitourinary sequelae in rectal cancer survivors and their impact on health-related quality of life: Outcome of a high-resolution population-based study. Surgery. 2019 Sep;166(3):327-335. doi: 10.1016/j.surg.2019.04.007. Epub 2019 Jun 14. PMID 31204071